CLINICAL TRIAL: NCT00169247
Title: Larynx Preservation With Induction Chemotherapy (Cisplatin, 5FU, Docetaxel) Followed by Radiotherapy Combined With Either Cisplatin or Cetuximab in Laryngopharyngeal Squamous Cell Carcinoma - A Randomised Phase II Study
Brief Title: Radiotherapy With Cisplatin Versus Radiotherapy With Cetuximab After Induction Chemotherapy for Larynx Preservation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Tumor Study Group Head and Neck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC-TREMPLIN
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Larynx Cancer; Hypopharynx Cancer
Keywords: larynx cancer; hypopharynx cancer; larynx preservation; concomitant radiochemotherapy; cisplatin; cetuximab; randomized trial
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Cetuximab; Cisplatin

INTERVENTIONS:
Drug: cetuximab
Drug: Cisplatin
Procedure: Radiotherapy 70 Gy, 35 fractions

SUMMARY:
Larynx preservation remains a very challenging approach in patients with larynx/pharynx cancer. A first attempt consisted of induction chemotherapy followed in good responders by irradiation. This approach allowed to preserve 60 % of the larynx without any significant difference in survival. The second attempt consisted of concurrent chemo-irradiation. This approach provided a higher larynx preservation rate but survival remained unchanged and mucosal toxicity was also higher. A third approach is currently under evaluation: induction chemotherapy followed by concurrent chemo-irradiation in good responders.

DETAILED DESCRIPTION:
At ASCO 2004 there were 3 major presentations issuing an increasing in survival:

* the update of the MACH-NC meta-analysis showed that actually only concurrent chemo-irradiation trials found a significantly improved survival (in particular the addition of cisplatinum alone to radiotherapy)
* the addition of docetaxel to the cisplatinum-5FU regimen (TPF) when compared with cisplatinum--5FU (PF)
* the addition of cetuximab to irradiation

On this basis we decided to carry-out a randomized phase II for previously untreated patients requiring a total laryngectomy:

All patients after a complete work-up including a CTscan will receive 3 cycles of TPF(T: 75 mg/m², P: 75 mg/m² and 5FU 750 mg/m²).

Patients with response over 50 % (endoscopy and CTscan) will be randomized to receive either irradiation (70 Gy) and cisplatinum (100 mg/m² on D1, D22 and D43) or irradiation (70 Gy) with cetuximab (loading dose of 400 mg followed by weekly 250 mg for a total of 8 cycles.

Patients with less than 50% decease in tumour volume after TPF, patients with residual or recurrent disease after either RT-CDDP or RT-cetuximab will get salvage total laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* Larynx or hypopharynx squamous cell carcinoma proven by histology, locally advanced, only eligible for surgery as total or sub-total (pharyngo-)laryngectomy
* Performance status 0-1
* Neutrophils >=1.5 x 109/l, Platelets count >=100 x 109/l, haemoglobin >=10 g/dl
* Total bilirubin <= 1.5 x upper reference range
* ASAT and ALAT <= 2.5 x upper reference range, Alkaline Phosphatases <= 5 x upper reference range
* Serum creatinine <= 120 µmol/l
* Weight loss < 10 % within last 3 months
* Written inform consent

Exclusion Criteria:

* Infiltrative transglottic tumor or clinical cartilage invasion
* Distant metastasis
* Previous chemotherapy or radiotherapy
* Contra-indication to chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2005-10; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
rate of laryngeal preservation

SECONDARY OUTCOMES:
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Lefebvre, Principal Investigator — Centre Oscar Lambret
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Centre René Gauducheau, Nantes
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Lefebvre JL, Pointreau Y, Rolland F, Alfonsi M, Baudoux A, Sire C, de Raucourt D, Malard O, Degardin M, Tuchais C, Blot E, Rives M, Reyt E, Tourani JM, Geoffrois L, Peyrade F, Guichard F, Chevalier D, Babin E, Lang P, Janot F, Calais G, Garaud P, Bardet E. Induction chemotherapy followed by either chemoradiotherapy or bioradiotherapy for larynx preservation: the TREMPLIN randomized phase II study. J Clin Oncol. 2013 Mar 1;31(7):853-9. doi: 10.1200/JCO.2012.42.3988. Epub 2013 Jan 22. PMID 23341517
- See also: Related Info — http://www.gettec.org